CLINICAL TRIAL: NCT02337556
Title: The DIVINE Study: DIetary Management of Glucose VarIability iN thE ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13.23.CLI
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Critically Ill Mechanically Ventilated Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Peptamen Bariatric
  Interventions: Other: Peptamen Bariatric
- Control Group (Active Comparator): Replete
  Interventions: Other: Replete

INTERVENTIONS:
Other: Peptamen Bariatric — Commercially available enteral diet
  Arms: Intervention Group
Other: Replete — Commercially available enteral diet
  Arms: Control Group

SUMMARY:
To compare the nutritional effect on blood glucose of two commercially available enteral diets in overweight or obese patients in the Intensive Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* New admit to the ICU and expected to remain in ICU 5 days
* Ventilator dependent up to 48 hours prior to admission to the study
* Requiring tube feeding enteral nutrition (EN) 5 days
* Expected to receive 50% of caloric needs within 72 hours
* Body Mass Index 26-45

Exclusion Criteria:

* Trauma patients
* Major surgery in past 30 days or planned for next 7 days
* Diabetes mellitus (DM) type 1
* Admitted with diagnosis of diabetic ketoacidosis as primary diagnosis
* Pregnant or lactating
* Non-functioning GI tract
* Use of parenteral nutrition in past 30 days
* Admitted with burns > 20% body surface area
* Traumatic brain injury
* Hemodynamic instability that prevents delivery of EN > 24hr
* Unable to access GI tract for feeding via tube, unable to receive EN
* Other contraindication to tube feeding
* Any other condition that would not allow patient to complete the study protocol
* Use of enteral formula at enrollment that cannot be changed to the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Glucose variability - Number of glycemic events outside the serum glucose range of 110-150 mg/dl | First seven days in the ICU
  Number of glycemic events outside the serum glucose range of 110-150 mg/dl

SECONDARY OUTCOMES:
Glucose variability - Number of glycemic events between 80-110 mg/dl and 150-180 mg/dl | First seven days in the ICU
  Number of glycemic events between 80-110 mg/dl and 150-180 mg/dl
Glucose variability - Number of episodes of hypoglycemia (glucose < 80 mg/dl) | First seven days in the ICU
  Number of episodes of hypoglycemia (glucose < 80 mg/dl)
Glucose variability - Number of episodes of hyperglycemia (glucose > 180 mg/dl) | First seven days in the ICU
  Number of episodes of hyperglycemia (glucose > 180 mg/dl)
Glucose variability - Average glucose levels | First seven days in the ICU
  Average glucose levels
Need for exogenous insulin administration | First seven days in the ICU
  Number of administrations, amount of insulin received, number of times insulin order adjusted, circulating C-peptide at baseline, day 3, 5 and 7
Need for exogenous glucose administration | First seven days in the ICU
  Number of times of administration and amount of glucose received
Nursing time | First seven days in the ICU
  Time required to monitor glucose levels and adjust insulin regimens in subset of patients studied

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Emory University Hospital, Atlanta, Georgia
  - University of Chicago Medicine, Chicago, Illinois
  - University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky
  - Regions Hospital, Saint Paul, Minnesota
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Queen's University, Kingston, Ontario, Canada